CLINICAL TRIAL: NCT05631223
Title: Use of Telemedicine to Address 'Off Target' Symptoms in Psoriatic Arthritis (PsA): Implementation of PsOWellTM in PsA
Brief Title: Use of Telemedicine to Address 'Off Target' Symptoms in Psoriatic Arthritis (PsA)
Acronym: PsOWell
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 851058
Record Dates: First submitted 2022-11-18; First posted 2022-11-30 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Psoriatic Arthritis
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — Telemedicine

STUDY DESIGN:
Intervention Model Description: This is a single-arm, multisite pilot study
Masking Description: As a pilot study to understand implementation barriers, assess feasibility, and effectiveness, this study is not blinded or randomized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional Telemedicine Arm (Experimental): Single Arm Intervention
  Interventions: Behavioral: Telemedicine

INTERVENTIONS:
Behavioral: Telemedicine — The intervention will consist of two structured telemedicine visits delivered between two routine office visits and conducted by providers (nurse practitioners and clinical nurse specialists).

SUMMARY:
This will be a single-arm interventional study to test the acceptability, feasibility, and effectiveness of structured telemedicine visits to encourage lifestyle changes that will improve quality of life, disease impact, and disease activity in patients with psoriatic arthritis (PsA).

DETAILED DESCRIPTION:
The proposed trial will be embedded within clinical care. This is a 2-year interventional trial that will enroll patients with active psoriatic arthritis despite stable therapy among three centers (the University of Pennsylvania, University of Utah, and University of Oxford). The intervention employs PsOWellTM, a program that trains clinicians to utilize motivational interviewing to help patients set goals and make lifestyle/behavior changes for holistic management of psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Population: Patients with Psoriatic Arthritis

  * Age 18-89.
  * Active symptoms of PsA as defined by a PsA Impact of Disease (PsAID) questionnaire score >4 (range 0-10, 4 is the patient acceptable symptom state) or a patient global assessment of greater than 4 (scale 0-10).
  * Patients should be stable on therapy (i.e., not planning to switch therapy at the current visit).
  * Meet CASPAR criteria.
  * Provision of signed and dated informed consent form.
  * Willingness to comply with all study procedures and availability for duration of the study.
  * Has access to a mobile phone or other mobile device.

Exclusion Criteria:

* Inability to provide informed consent.
* Plan to change systemic treatment for psoriasis or PsA in the next 4-8 weeks.
* PsAID score ≤4

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Estimated)
Dates: Start 2023-03-10 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Acceptability | 4 Months
  Patient satisfaction as assessed by Acceptability of Intervention Measure (AIM). The range of this measure is 4-20 where higher scores indicate greater acceptability and satisfaction
Effectiveness | 4 Months
  Effectiveness as measured by the Psoriatic Arthritis Impact of Disease 12-item questionnaire (PSAID-12) Survey. The range of the final PsAID-12 value is 0-10 where higher figures indicate worse status.
Minimal Disease Activity | 4 Months
  Minimal Disease Activity (MDA) Composite Score. MDA measures the state of the patient's disease activity. Achievement of MDA means attaining 5/7 of the following: Swollen Joint Count (SJC) ≤1, Tender Joint Count (TJC) ≤1, Enthesitis ≤1, Psoriasis Body Surface Area (BSA) ≤3%, Patient Global Assessment ≤ 20 (0-100), Patient Pain ≤ 20 (0-100), and Health Assessment Questionnaire (HAQ) <0.05 (0-3). It is a patient-reported and physician-assessed outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Alexis Ogdie-Beatty, MD, Principal Investigator — University of Pennsylvania
Locations (2):
- United States (2):
  - University Of Pennsylvania, Philadelphia, Pennsylvania
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No
Fully de-identified datasets will be shared with requesting parties after manuscript publication and following submission of a protocol by the requesting party and approval by the study investigators.